CLINICAL TRIAL: NCT02975843
Title: Open Label, Uncontrolled, Non-randomized, Single Dose, Scintigraphic Study to Investigate Lung Deposition of Inhaled 99mTc Radiolabelled CHF5993 pMDI in Healthy Volunteers, Asthmatic and COPD Patients
Brief Title: Lung Deposition of Beclometasone Dipropionate/Formoterol Fumarate/Glycopyrronium Bromide Administered Via pMDI in Healthy, Asthmatic and COPD Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCD-05993AA1-15; 2016-001088-35 (EudraCT Number)
Record Dates: First submitted 2016-11-15; First posted 2016-11-29 (Estimated); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Chronic Obstructive Pulmonary Disease; Asthma
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma | interventions — Beclomethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CHF5993 (Experimental): 99mTc Radiolabelled Beclometasone dipropionate/Formoterol Fumarate/Glycopyrronium Bromide administered via pMDI
  Interventions: Drug: Beclometasone dipropionate/Formoterol Fumarate/Glycopyrronium

INTERVENTIONS:
Drug: Beclometasone dipropionate/Formoterol Fumarate/Glycopyrronium — single inhalation of 99mTc radiolabelled CHF 5993 pMDI (4 puffs for a total dose of: Beclometasone diproprionate (BDP) 400 μg, Formoterol fumarate (FF) 24 μg, Glycopirronium bromide (GB) 50 μg)
  Other Names: CHF5993 pMDI

SUMMARY:
The purpose of this study is to investigate the lung deposition and distribution pattern of Beclometasone dipropionate/Formoterol Fumarate/Glycopyrronium Bromide using a Gamma-scintigraphic technique after inhalation of a single dose of 99mTc radiolabelled CHF 5993 Administered via pMDI in healthy volunteers, asthmatic and COPD patients.

ELIGIBILITY:
Inclusion Criteria for all subjects:

1. Subject's written informed consent obtained prior to any study-related procedure
2. Body mass index (BMI) between 18 and 32 kg/m2
3. Ability to understand the study procedures and the risks involved and ability to be trained to use the devices correctly at screening and pre-dose.
4. Normal vital signs (Diastolic BP 60-90 mmHg, Systolic BP 90-140 mmHg or 90-150 if >45 yrs) at screening and pre-dose.
5. 12-lead digitalised ECG considered as normal: 60 ≤ heart rate ≤ 100 bpm, 120 ms ≤ PR ≤210 ms, QRS ≤ 120 ms, QTcF ≤ 450 ms (male) and ≤ 470 ms (female) at screening and pre-dose
6. Males fulfilling one of the following criteria:

   1. Males with non-pregnant Women of childbearing potential (WOCBP) partners: they and/or their partner of childbearing potential must be willing to use a highly effective birth control method in addition to the male condom from the signature of the informed consent and until 90 days after the follow-up visit. Subjects must not donate sperm during the study and for 90 days after the follow-up visit or
   2. Males with pregnant WOCBP partner: they must be willing to use male contraception (condom) from the signature of the informed consent and until 90 days after the follow-up visit. Subjects must not donate sperm during the study and for 90 days after the follow-up visit or
   3. Non-fertile male subjects (contraception is not required in this case) or
   4. Males with partner not of childbearing potential (contraception is not required in this case).
7. WOCBP fulfilling one of the following criteria:

   1. WOCBP with fertile male partners: they and/or their partner must be willing to use a highly effective birth control method with low user dependency from the signature of the informed consent and until 30 days after the follow-up visit or
   2. WOCBP with non-fertile male partners (contraception is not required in this case).
8. Female patients of non-childbearing potential defined as physiologically incapable of becoming pregnant (i.e. post-menopausal or permanently sterile). Tubal ligation or partial surgical interventions are not acceptable. If indicated, as per investigator's request, post-menopausal status may be confirmed by follicle-stimulating hormone levels (according to local laboratory ranges)

   Additional Inclusion criteria for Healthy /volunteers and Asthmatic patients:
9. Males and females aged 18-55
10. Non- or Ex-smokers who smoked < 5 pack years (pack-years = number of cigarette packs per day times the number of years) and stopped smoking > 1 year

    Additional Inclusion Criteria only for Healthy volunteers:
11. Lung function within normal limits: FEV1 ≥ 80% of predicted (according to the Global Lung Function Initiative, ERS Task Force Lung Function Reference Vales) and FEV1/FVC ratio > 0.70 at screening

    Additional Inclusion Criteria only for Asthmatic patients:
12. Pre-bronchodilator 60% ≤ FEV1 ≤ 80% of predicted (according to the Global Lung Function Initiative, ERS Task Force Lung Function Reference Vales) and FEV1/FVC ratio > 0.70 at screening. If this criterion is not met at Screening, the test can be repeated once before Day -1.
13. Positive reversibility test as defined by an increase in FEV1 ≥ 12% and at least 200 ml compared to the initial value 20-30 minutes after inhalation of 400 μg Salbutamol at screening. If this criterion is not met at Screening, the test can be repeated once before Day -1.

    Additional Inclusion Criteria only for COPD patients:
14. Males and females aged 40-75
15. Current or ex- smokers (stopped smoking > 1 year ) minimum smoking history of 10 pack-years (packyears = number of cigarette packs per day times the number of years)
16. 30% ≤ FEV1 < 50% of predicted and FEV1/FVC < 0.70 after inhalation of 400 μg Salbutamol. If this criterion is not met at Screening, the test can be repeated once before Day -1.

Exclusion Criteria for all subjects:

1. Pregnant or lactating women
2. Documented history of drug abuse (within 12 months before screening) and/or positive urine drug test at screening and/or at treatment period
3. History of hypersensitivity to M3 Antagonists, β2-agonist, corticosteroids or any of the excipients contained in any of the formulations used in the trial;
4. Any clinically relevant abnormal laboratory value at screening suggesting an unknown disease and requiring further clinical investigation or which may impact the safety of the subject or the evaluation of the result of the study according to the investigator's judgment
5. Clinically relevant and uncontrolled hepatic, gastrointestinal, renal, genitourinary, endocrine, metabolic neurologic, or psychiatric disorder that may interfere with successful completion of this protocol
6. Serology at the screening positive to HIV1 or HIV2 and positive results for Hepatitis which indicates acute or chronic Hepatitis B (i.e. positive HB surface antigen HBsAg positive and/or positive HB core antibody anti-HBc) or Hepatitis C (HCV antibody);
7. Subjects with history of sustained and non-sustained cardiac arrhythmias (ECG demonstrated) and subjects with a family history of sudden cardiac death
8. Subjects who have cardiovascular condition such as, but not limited to unstable ischemic heart disease, NYHA Class III/IV left ventricular failure, acute ischemic heart disease in the last year prior to study screening, which may impact the safety of the subject or the evaluation of the result of the study according to the investigator's judgment
9. Medical diagnosis of narrow-angle glaucoma, prostatic hypertrophy or bladder neck obstruction that in the opinion of the investigator would prevent use of anticholinergic agents"
10. Significant blood loss ≥ 400 ml within 3 months prior screening and between screening and Day 1;
11. Participation in another clinical trial with an investigational drug in the previous 3 months before the administration of the study drug; a longer and more appropriate time could be considered by the principal investigator based on the elimination of the half-life and/or long term toxicity of the previous investigational drug;
12. Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 1999, shall participate in the study.
13. Unsuitable veins for repeated venipuncture
14. Any not allowed concomitant medication

    Additional Exclusion criteria for Healthy volunteers and Asthmatic patients:
15. Current use of any nicotine or nicotine replacement product

    Additional Exclusion criteria for Asthmatic and COPD patients:
16. Use of systemic steroids in the 4 weeks prior to screening and between screening and Day 1 (injectable depot steroids 6 weeks)
17. Life-threatening/unstable respiratory status including upper or lower respiratory tract infection, within the previous 30 days before screening and between screening and Day 1
18. Requirement for continuous oxygen therapy (supplemental oxygen not exceeding 2 l/min, at night only and/or during exercise is allowed)

    Additional Exclusion criteria only for asthmatic patients:
19. Change in dose or type of any medications for asthma within 4 weeks prior to the screening visit
20. Asthma exacerbation within the 4 weeks prior screening and between screening and Day 1
21. History of COPD or any chronic respiratory disease other than Asthma

    Additional Exclusion criteria only for COPD patients:
22. Change in dose or type of any medications for COPD within 4 weeks prior to the screening visit
23. COPD exacerbation within the 4 weeks prior screening and between screening and Day 1
24. History of asthma or any chronic respiratory disease other than COPD

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-11-21 (Actual); Primary Completion 2017-03-21 (Actual); Study Completion 2017-04-11 (Actual)

PRIMARY OUTCOMES:
Intrapulmonary Lung deposition expressed as % of nominal dose | Immediately after dosing
  Calculated using the individual Gamma camera images

SECONDARY OUTCOMES:
Distribution of lung deposition | Immediately after dosing
  Calculated using the individual Gamma camera images
Extrathoracic deposition | Immediately after dosing
  Calculated using the individual Gamma camera images
Exhaled activity | Immediately after dosing
  Calculated using the individual Gamma camera images
BDP/B17MP, Formoterol, and GB Area under curve (AUC) 0-t | the area under the plasma concentration-time curve from 0 to the last quantifiable concentration. Over 24h
  Calculated through plasma samples for PK evaluation
BDP/B17MP, Formoterol, and GB Area under curve (AUC) 0-30min | area under the plasma concentration-time curve from 0 to 30 min post-dose
  Calculated through plasma samples for PK evaluation
BDP/B17MP, Formoterol, and GB area under the curve (AUC) 0-∞ | area under the curve extrapolated to infinity over 24h
  Calculated through plasma samples for PK evaluation
BDP/B17MP, Formoterol, and GB Peak Plasma Concentration (Cmax) | the value of the maximum plasma concentration will be obtained directly from the experimental data without interpolation. Over 24h
  Calculated through plasma samples for PK evaluation
BDP/B17MP, Formoterol, and GB tmax | time of the maximum plasma concentration will be obtained directly from the experimental data without interpolation. Over 24h
  Calculated through plasma samples for PK evaluation
BDP/B17MP, Formoterol, and GB t½ | the terminal (apparent elimination) half-life over 24h
  Calculated through plasma samples for PK evaluation
lung function assessment | Over 24 h post dose
  Calculated using spirometry